CLINICAL TRIAL: NCT04087629
Title: Post-marketing Surveillance of StrataCTX® Flexible Wound Dressing for Use as a Steroid Sparing Agent
Brief Title: StrataCTX® as a Steroid Sparing Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Larisa Geskin, MD, Principal Investigator, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAR6582
Record Dates: First submitted 2019-02-01; First posted 2019-09-12 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: CTCL
Keywords: CTCL; topical steroids; StrataCTX®; cutaneous; steroid sparing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CTCL group (Experimental): Patients with CTCL being treated with mechlorethamine gel will receive StrataCTX® gel.
  Interventions: Device: StrataCTX® gel

INTERVENTIONS:
Device: StrataCTX® gel — Gel forming flexible wound dressing for the prevention and treatment of radiation dermatitis

SUMMARY:
The purpose is to determine if StrataCTX® can be used as a steroid sparing agent for the treatment of cutaneous reactions related to, cutaneous T Cell lymphoma (CTCL) and chemotherapy/immunotherapy treatments than the current standard treatment - topical steroids - in people who are receiving treatment for CTCL, or chemotherapy/immunotherapy for solid/hematologic malignancies. Subjects will have CTCL and are being treated with topical steroids, or being treated with chemotherapy/immunotherapy for another condition and have had cutaneous reactions that have warranted initiation of topical steroids.

DETAILED DESCRIPTION:
Topical steroids are the mainstays of treatment for many cutaneous reactions and disorders. Steroids are known to cause many side effects and few effective pharmacologic alternatives exist. Contact dermatitis is observed in 56% of patients with cutaneous T-cell lymphoma (CTCL) being treated with topical mechlorethamine gel. This usually requires chronic treatment with mid-to high-potency steroids. Numerous chemo/immunotherapies are associated with cutaneous reactions including paronychia, hand and foot syndrome, and acneiform rash. Skin toxicity often requires dose reduction of cancer therapies and a variety of skin directed therapies including topical antibiotics and topical steroids. Cutaneous reactions are often the earliest manifestation of acute graft versus host disease. Skin manifestations can be debilitating and treatment usually requires high potency topical steroids. Additional therapies are needed for the treatment of disorders that rely on topical steroids.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ability to sign informed consent document
* Patient with a diagnosis of CTCL who have contact dermatitis to topical mechlorethamine gel
* Patients with a diagnosis of CTCL who have intractable pruritis
* Patients with a diagnosis of CTCL who rely heavily on topical steroids for symptomatic relief
* Patients on chemo/immunotherapy with drug induced rash

Exclusion Criteria:

* Patients currently undergoing radiotherapy
* Patients currently receiving oral steroids
* Patients who are unable to apply topical medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Pruritus Visual Analogue Scale (VAS) Score | Screening through 3 months
  The primary objective of this study is to determine whether StrataCTX® gel is effective as a supportive therapy for cutaneous reactions treated with topical steroids as the standard of care. This objective will be measured by the Pruritus Visual Analogue Scale, which measures self-reported itching on a scale of 0 (no itching) (better outcome) to 10 (worst imaginable itch).

SECONDARY OUTCOMES:
Change in SKINDEX-16 Quality of Life (QOL) Score | Screening through 3 months
  Another objective is to determine if StrataCTX® will improve patient quality of life secondary to symptomatic improvement through the use of the Skindex 16 QOL (a dermatologic quality-of-life instrument) , which is a validated measure where participants self-report from 1 (never) - 5 (all the time) how each of 30 statements describes participants feelings related to their skin condition. All responses are transformed to a linear scale of 100, varying from 0 (no effect) (better outcome) to 100 (effect experienced all the time).
Change in the Rate of Primary Skin Reactions | Screening through 3 months
  Change in the rate of primary skin reactions in participants between the topical steroid treatment period, compared to the StrataCTX® gel period as evaluated in screening visits.
Change in Topical Steroid Use | Day 30 through 3 months
  Change in topical steroid use during the StrataCTX® gel period as reported daily in patient diaries with time, date, and location of topical steroid application.

CONTACTS AND LOCATIONS:
Overall Officials: Larisa J. Geskin, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Clinical Endpoints/ individual patient data (IPD) will be assessed based on analysis of photos and evaluation of survey data, including scores from Pruritis VAS and Skindex-16 QOL scales. The scores during topical steroid treatment period will be compared to the scores during the StrataCTX® gel treatment period. Safety endpoints will be evaluated based on report of product related adverse events and subsequent study product interruption.

REFERENCES:
- See also: StrataCTX Informational Pamphlet — https://stratactx.com/wp-content/uploads/2020/10/StrataCTX-Detail-Aid-Master-Language-English-CT-ML-007-2-0619-4.pdf
- See also: StrataCTX FAQS — https://stratactx.com/faqs/